CLINICAL TRIAL: NCT00320892
Title: "Death Rattle" - A Double Blind, Randomly Controlled, Crossover Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting appropriate participants to the study
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Pesach Shvartzman, Head Family Medicine Department, Soroka University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOR416506CTIL
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Noise; Death
Keywords: Death Rattle; Noise level; Primary Care
MeSH Terms: conditions — Death | interventions — Atropine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Atropine Sulphate 1% ophthalmic drops — Atropine Sulphate 1% ophthalmic drops will be used, by Fisher Pharmaceutical Labs, at a dose of 2 drops per administration

SUMMARY:
Dying patients are often unable to clear secretions from their large airways, resulting in noisy breathing usually described as "death rattle." While there is no evidence that patients find this condition disturbing, the noises may be disturbing to the patient's visitors and caregivers who may fear that the patient is choking to death.

In Israel none of the pharmaceutical drugs listed in the literature exist. Thus, Atropine drops which have been noted in the literature as being used, though according to our knowledge no evidence of clinical trials using sublingual Atropine were conducted.

The study is designed as a randomly controlled, double blind crossover trial. The patient will serve as control for himself, as crossover between placebo and drug (randomly chosen) will take place. The administrator of the drug will be blinded to the medication, each time randomly beginning with a different drug (placebo or Atropine).

We will evaluate Atropine Sulphate 1% ophthalmic drops effect on 33 patients using a noise score scale of 0-3. Noise scores will be taken at the start; 30 min after drug/placebo administration and every hour thereafter. After 4-hours crossover will take place and evaluation will follow the same protocol.

ELIGIBILITY:
Inclusion Criteria:

* : Patients belonging to Home Palliative Care Unit of Clalit Health Services - Southern District, and the Oncology Department of Soroka University Medical Center and suffering from "death rattle" will be recruited for the study.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Noise Level | 8 hours
  30 min after drug administration; and hourly after the initial administration. if needed a repeat dose will be given and the noise score will be evaluated at 30 min; and hourly thereafter. The repeat dose will be left to the nurses' discretion if they thought the rattle to be unacceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Pesach Shvartzman, Study Chair — Ben-Gurion University of the Negev
Locations (1):
- Ben-Gurion University of the Negev, Sial Research Center for Family Medicine and Primary Care, Beersheba, Israel